CLINICAL TRIAL: NCT03570242
Title: Effect of Whole-body Electromyostimulation Combined With Individualized Nutritional Support on Patients With Gynecological Cancer Undergoing Curative and Palliative Treatment
Brief Title: WB-EMS and Individualized Nutritional Support in Gynecological Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Gyn EMS
Record Dates: First submitted 2018-06-01; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Gynecologic Cancer; Cachexia
Keywords: gynecologic cancer; WB-EMS; whole-body electromyostimulation; nutrition; protein; exercise; cancer cachexia
MeSH Terms: conditions — Cachexia; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (palliative treatment) (No Intervention): "usual care" control group (includes patients undergoing palliative Treatment) receives individualized nutritional support (dietary advices: daily protein intake1,2 - 1,5 g/kg bodyweight)
- WB-EMS group (palliative treatment) (Experimental): physical exercise group (includes patients undergoing palliative Treatment) receives regular WB-EMS training (2 EMS trainings per week; each session for 20 min)
  + individualized nutritional support (dietary advices: daily protein intake 1,2-1,5 g/kg bodyweight)
  Interventions: Other: Whole-Body Electromyostimulation (WB-EMS)
- Control group (curative treatment) (No Intervention): "usual care" control group (includes patients undergoing curative treatment 3-4 weeks before surgery) receives individualized nutritional support (dietary advices: daily protein intake1,2 - 1,5 g/kg bodyweight)
- WB-EMS group (curative treatment) (Experimental): physical exercise group (includes patients undergoing adjuvant treatment 3-4 weeks before surgery) receives regular WB-EMS training (2 EMS trainings per week; each session for 20 min)
  + individualized nutritional support (dietary advices: daily protein intake 1,2-1,5 g/kg bodyweight)
  Interventions: Other: Whole-Body Electromyostimulation (WB-EMS)

INTERVENTIONS:
Other: Whole-Body Electromyostimulation (WB-EMS) — WB-EMS training is performed 2x/week for 12 weeks; Stimulation protocol: Frequency of 85 Hz, pulse duration of 0.35 ms, stimulation period of 6 sec, resting period of 4 sec; supervised by certified training instructors/physiotherapists participants perform simple exercises during the stimulation period following a video tutorial
  Arms: WB-EMS group (curative treatment); WB-EMS group (palliative treatment)

SUMMARY:
This study evaluates the effects of a 12-week whole-body electromyostimulation (WB-EMS) training combined with individualized nutritional support on body composition, muscle strength and function, quality of life, fatigue and Inflammatory status on patients with gynecological cancer undergoing palliative anti-cancer Treatment. Furthermore, this study assesses the effect of this combined therapeutic approach within a 3 to 4-week pre-operative study Intervention on the period of hospitalization in gynecological patients undergoing curative anti-cancer Treatment.

ELIGIBILITY:
Inclusion Criteria:

* female patients with gynecological cancer undergoing palliative or curative treatment
* 18 years and older
* ECOG status > 2

Exclusion Criteria:

* simultaneous participation in other nutritional or exercise intervention Trials or in the past 6 months
* acute cardiovascular events
* use of anabolic medications
* epilepsy
* severe neurological diseases
* skin lesions in the area of electrodes
* energy active metals in body
* pregnancy
* acute vein thrombosis
* rheumatic diseases
* pregnant and nursing women
* psychiatric disorders with doubts about legal and cognitive capacity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Skeletal muscle mass | 12 weeks (palliative treatment), 3-4 weeks (curative treatment)
  Skeletal muscle mass assessed by bioelectrical impedance analysis (in kg)
Period of hospitalization | 3-4 week (curative treatment)
  Days of Hospital stay after curative surgery

SECONDARY OUTCOMES:
Physical function - Isometric muscle strength | 12 weeks (palliative treatment), 3-4 weeks (curative treatment)
  Hand grip strength assessed by hand dynamometer (in kg)
Physical function - Endurance | 12 weeks (palliative treatment), 3-4 weeks (curative treatment)
  Six-minute-walk test (walking distance in m)
Physical function - Lower limb strength | 12 weeks (palliative treatment), 3-4 weeks (curative treatment)
  30 second sit-to-stand test (number of sit-to-stand cycles)
Patient-reported performance status | 12 weeks (palliative treatment), 3-4 weeks (curative treatment), Total Score ranges from 0-100 with a higher score indicating better performance status
  Karnofsky index
Patient-reported Quality of Life (QoL) | 12 weeks (palliative treatment), 3-4 weeks (curative treatment)
  European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC QLQ - C30); Total score ranges from 0-100 with a higher score indicating better functioning/Quality of life or higher symptom burden
Patient-reported Fatigue | 12 weeks (palliative treatment), 3-4 weeks (curative treatment)
  FACIT-Fatigue scale; Total score ranges from 0-52 with a higher score indicating better Quality of life/less fatigue
Pain score | 12 weeks (palliative treatment), 3-4 weeks (curative treatment)
  Visual Analogue Scale (VAS); Total score ranges from 0-10 with a higher score indicating higher pain
Depression score | 12 weeks (palliative treatment), 3-4 weeks (curative treatment)
  Beck Depression Inventory (BDI); Total score ranges from 0-63 with higher score indicating higher depression
Gastrointestinal toxicity of chemotherapy | 12 weeks (palliative treatment), 3-4 weeks (curative treatment)
  Number of participants with treatment-related adverse events of gastrointestinal toxicity as assessed by CTCAE v4.0
Physical activity | 12 weeks (palliative treatment), 3-4 weeks (curative treatment)
  International Physical Activity Questionnaire (IPAQ); Higher score indicates higher physical acitivity level
Inflammatory status | 12 weeks (palliative treatment), 3-4 weeks (curative treatment)
  Analysis of serum C-reactive protein (CRP) and albumin concentrations

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine 1, Hector Center for Nutrition, Exercise and Sports, Friedrich-Alexander-University Erlangen-Nuremberg, Erlangen, Germany